CLINICAL TRIAL: NCT04665817
Title: Diagnostic Accuracy of CCTA-derived Versus AngiogRaphy-dErived QuantitativE Flow Ratio Study
Brief Title: Diagnostic Accuracy of CCTA-derived Versus AngiogRaphy-dErived QuantitativE Flow Ratio (CAREER) Study
Acronym: CAREER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanghai Jiao Tong University -Pulse Medical Imaging Technology Joint Lab (Unknown)
Responsible Party: Principal Investigator, Zhijun Bao, Huadong Hospital, Department of Cardiology, Fudan University
Other Study IDs: Huadong Hospital
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Coronary Stenosis; Hemodynamics; Coronary Artery Disease; Coronary Computed Tomography Angiography
Keywords: coronary stenosis; coronary computed tomography angiography; hemodynamics; CT-QFR; QFR
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT-QFR — CT-QFR is a novel method for evaluating the functional significance of coronary stenosis. It is calculated by coronary computed tomographic angiography images.
  Other Names: Fast Computational Approach to Derive Fractional Flow Reserve From Coronary CT Angiography
Diagnostic Test: QFR — QFR is a novel method for evaluating the functional significance of coronary stenosis by calculation of the pressure drop in the vessel based on two. angiographic projections.
  Other Names: Quantitative Flow Ratio
Diagnostic Test: FFR — FFR measured by pressure wire is the gold standard for evaluating the functional significance of coronary stenosis.
  Other Names: Fraction Flow Reserve

SUMMARY:
To perform CT-QFR, invasive coronary angiography, FFR, and QFR tests on patients with moderate coronary stenosis after coronary CTA examination. Use FFR as a reference to verify the diagnostic performance of CT-QFR, and compare it with QFR.

DETAILED DESCRIPTION:
This study is a prospective and single-center trial in China.It intends to enroll 216 patients with coronary artery disease whose coronary artery is determined to be 30-90% stenosis after coronary CT scan. CT image data will be imported for CT-QFR detection and undergo coronary angiography within 30 days. Quantitative analysis of coronary angiography (QCA) was performed with the degree of coronary stenosis. FFR and QFR were detected during the operation. Use FFR as a reference standard to verify the diagnostic performance of CT-QFR and QFR. The primary endpoint is the diagnostic accuracy of CT-QFR in identifying hemodynamically significant coronary stenosis with FFR as the reference standard. Major secondary endpoint is the non-inferiority of CT-QFR compared with QFR in the patients without extensively calcified lesions. The completion of the project will provide patients with a practical non-invasive assessment method of coronary heart disease which provides the best treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Coronary CT angiography indicates that >= 1 stenosis with percent diameter stenosis between 30%-90% in a vessel >= 2mm.
2. The invasive coronary angiography should be less than 30 days after the coronary CT angiography.

Exclusion Criteria:

1. The target lesion has received coronary stent implantation or coronary artery bypass graft.
2. Target lesion involves myocardial bridge.
3. Severe heart failure (NYHA ≥III).
4. Renal function is seriously damaged (eGFR<30 ml/min/1.73m2).
5. Those who are contraindicated to use contrast agents, beta blockers, nitrates or adenosine drugs.
6. Acute myocardial infarction within 1 month.
7. The image quality of CTA or coronary angiography cannot be assessed.
8. Any factors that affect the image quality of coronary CTA and coronary angiography, such as frequent premature contractions, atrial fibrillation, etc.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled patients are adults with suspected CAD who underwent clinically indicated ICA after CT which indicates moderate coronary artery stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of CT-QFR | 1.5 year
  Diagnostic accuracy of on-site CT-QFR in identifying physiologically significant coronary artery stenosis, using FFR as the reference standard.
  Presence of hemodynamically-significant coronary artery stenosis : FFR <= 0.80.

SECONDARY OUTCOMES:
Comparision between CT-QFR and QFR | 1.5 year
  Use FFR as a reference standard to validate the non-inferiority of CT-QFR compared with QFR in the vessels without extensively calcified lesions defined by the combination of a cross-sectional calcium arc >90° and a thickness >1.5 mm. For CT-QFR, QFR and FFR evaluations, vessels with <=0.80 are regarded as having hemodynamically significant CAD.
Other common measures of diagnostic performance of CT-QFR | 1.5 year
  Other common measures of diagnostic performance of CT-QFR, including sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) at the patient level compared with FFR as the reference standard.
  Presence of hemodynamically-significant coronary artery stenosis : FFR <= 0.80.
Correlation between CT-QFR and FFR | 1.5 year
  Pearson correlation or spearman's correlation will be used to quantify the correlations between CT-QFR and FFR. Agreements between CT-QFR and FFR will be assessed by Bland-Altman plot.
  The correlation coefficient r=0-0.2 represents very weak or no correlation. 0.2-0.4 represents weak correlation. 0.4-0.6 represents moderate correlation. 0.6-0.8 represents strong correlation. 0.8-1.0 represents very strong correlation.
The comparison between CT-QFR, CCTA-derived percent diameter stenosis (CTA-DS%) and QCA-derived DS% | 1.5 year
  The comparison of the discrimination ability between CT-QFR, CCTA-derived percent diameter stenosis (CTA-DS%), and QCA-derived DS% for identifying physiologically significant stenosis with FFR as the reference standard.
  Presence of hemodynamically-significant coronary artery stenosis : FFR <= 0.80.

CONTACTS AND LOCATIONS:
Overall Officials: Xinkai Qu, MD,PhD, Principal Investigator — Huadong Hospital, Department of Cardiology; Tingwen Weng, MD, Principal Investigator — Huadong Hospital, Department of Cardiology
Locations (1):
- Xinkai Qu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weng T, Ding D, Li G, Guan S, Han W, Gan Q, Li M, Qi L, Li C, Chen Y, Zhang L, Li T, Chang X, Chen Y, Wijns W, Qu X, Tu S. Accuracy of coronary computed tomography angiography-derived quantitative flow ratio for onsite assessment of coronary lesions. EuroIntervention. 2024 Oct 21;20(20):e1288-e1297. doi: 10.4244/EIJ-D-24-00336. PMID 39432253
- [Derived] Weng T, Gan Q, Li Z, Guan S, Han W, Zhai X, Li M, Qi L, Li C, Chen Y, Zhang L, Chang X, Tu S, Qu X. Diagnostic accuracy of CCTA-derived versus angiography-derived quantitative flow ratio (CAREER) study: a prospective study protocol. BMJ Open. 2022 Jun 23;12(6):e055481. doi: 10.1136/bmjopen-2021-055481. PMID 35738652